CLINICAL TRIAL: NCT02128867
Title: Influence of Bouncing, Assisted Autogenic Drainage (AAD) and Bouncing and AAD (BAAD) on Gastro-oesophageal Reflux ( GOR ), Oxygen Saturation (SaO2) and Heart Rate in Infants From 0 to 12 Months
Brief Title: Safety Study of Airway Clearance Techniques in Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Filip Van Ginderdeuren, PT, Drs., Vrije Universiteit Brussel
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVG001
Record Dates: First submitted 2014-04-23; First posted 2014-05-01 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Gastro-esophageal Reflux
Keywords: gastro-esophageal reflux; GOR; GER; airway clearance techniques
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Assisted Autogenic Drainage (AAD) (Experimental): airway clearance technique for infants :Assisted Autogenic Drainage
  Interventions: Other: Assisted Autogenic Drainage (AAD)
- bouncing and AAD (Experimental): airway clearance technique for infants : bouncing combined with AAD
  Interventions: Other: bouncing and AAD
- bouncing (Experimental): bouncing . intervention to relax the infant
  Interventions: Other: bouncing

INTERVENTIONS:
Other: Assisted Autogenic Drainage (AAD)
  Arms: Assisted Autogenic Drainage (AAD)
Other: bouncing and AAD
  Arms: bouncing and AAD
Other: bouncing
  Arms: bouncing

SUMMARY:
The purpose of this study is to determine whether three airway clearance techniques ( Bouncing, Assisted Autogenic Drainage ( AAD) and bouncing and AAD) provoke or aggravate gastro-esophageal reflux in infants under the age of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* infants < 1 year
* acid reflux monitoring

Exclusion Criteria:

* gestational age <24 w
* anti-reflux medication
* Nissen fundoplication
* no parental consent

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZBrussel, Jette, Brussels Capital, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Assisted Autogenic Drainage (AAD): airway clearance technique for infants :Assisted Autogenic Drainage
  Assisted Autogenic Drainage (AAD)
- Bouncing Combined With AAD: airway clearance technique for infants : bouncing combined with AAD
  bouncing combined with AAD
- Bouncing: bouncing as control group. intervention to relax the infant
  bouncing
Period: Overall Study
Arm/Group | Assisted Autogenic Drainage (AAD) | Bouncing Combined With AAD | Bouncing
Started | 53 | 52 | 54
Completed | 50 | 50 | 50
Not Completed | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Bouncing: bouncing . intervention to relax the infant
  bouncing
- Total: Total of all reporting groups
Arm/Group | Assisted Autogenic Drainage (AAD) | Bouncing Combined With AAD | Bouncing | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 50 | 150
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 22 | 69
  Male | 26 | 27 | 28 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Refluxes
Description: number of refluxes will be counted over a period of 15 minutes ( treatment time )
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: number of refluxes
Arm/Group | Assisted Autogenic Drainage (AAD) | Bouncing Combined With AAD | Bouncing
Number analyzed (Participants) | 50 | 50 | 50
number of refluxes | 0.48 (1.36) | 1.14 (2.55) | 1.62 (3.8)

2. Secondary Outcome: Duration of Reflux Episodes
Description: duration of reflux episodes will be measured during 15 min of treatment time
Time Frame: 15 minutes
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Heartrate
Description: heartrate will be measured during 15 min of treatment time
Time Frame: 15 minutes
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Sa02
Description: SaO2 will be measured during 15 minutes of treatment time
Time Frame: 15 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Assisted Autogenic Drainage (AAD) | Bouncing Combined With AAD | Bouncing
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/54
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No